CLINICAL TRIAL: NCT05293847
Title: Effects Of An Postural Based Telerehabilitation On Posture, Energy Consumption, and Performance In Mechanic Neck Pain
Brief Title: Postural Based Telerehabilitation in Mechanic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Director, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-80
Record Dates: First submitted 2022-03-08; First posted 2022-03-24 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Neck Pain; Telerehabilitation; Postural; Defect
Keywords: neck pain; telerahabilitation; posture
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Pre and post-intervention evaluations were compared in this study.
Masking Description: Individuals who perform telerehabilitation applications and evaluate the results are different.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation exercises (Experimental): Exercises about postural structures on the cervical and thoracal region. Bilateral pectoral stretching, chin tack exercises, cervical isotonic exercises, stretching of the upper trapezius and longus Colli, scapular region strengthening, shoulder capsular stretching, Wand exercises for 12 weeks and 3 times a week.
  Interventions: Behavioral: Telerehabilitation exercises and postural skills

INTERVENTIONS:
Behavioral: Telerehabilitation exercises and postural skills — 12 week based postural exercises and skills were applied to participants. The exercises were done 3 times a week. The exercises about cervical and thoracal region strengthening and stretching of muscles and structures.

SUMMARY:
It has been reported that staying in the same posture for a long time causes musculoskeletal system problems, and the use of mobile phones and other electronic devices continuously, especially in the internet age, causes postural problems in many people. Physiotherapy applications including strengthening, stretching, yoga, pain-oriented applications, and behavioral treatments are performed for an ideal posture to regulate postural problems. When the literature is examined, it has been seen that the studies carried out after the Covid 19 pandemic have developed especially in the direction of telerehabilitation, but there is a need for studies showing the effect of exercise applications developed for individuals with mechanical neck pain. This study was conducted to investigate the effect of 12-week telerehabilitation on posture, energy consumption, and performance in individuals with mechanical neck pain.

DETAILED DESCRIPTION:
This cross-sectional study was conducted at the Faculty of Physiotherapy and Rehabilitation, University of Health Sciences. All evaluations were performed in the university physiotherapy laboratories. All of the participants were informed about the study and provided written informed consent. This study was performed in accordance with the 1964 Helsinki declaration, its later amendments.110 people over the age of 18 were included in the study. Posture-oriented exercises were applied online 3 times a week for 12 weeks. Postural measurements, performance, and energy consumption levels were determined for each participant before and after the intervention. Craniovertebral angle and shoulder angle were measured with a smartphone application and muscle shortness was measured with clinical tests among postural measurements. Performance measurement was evaluated with the 6-minute walking test, and energy consumption was evaluated with the Physiological Cost Index. Individuals diagnosed with mechanical neck pain who applied to the university's wellness center for exercise between September 2021 and December 2021 were determined by physiotherapists who are experts in their fields. A cross-sectional selection of 110 individuals met the inclusion criteria. This study was conducted with assessments made before and after posture-based telerehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were being aged 18 years or over,
* Volunteering to take part in the study,
* Being a student of online education,
* without a history of any neurological or orthopedic problem,
* with resting neck pain (as measured by the Visual Analogue Scale) lasting ≤30 days and that is aggravated by movement without extending distal to the shoulders.

Exclusion Criteria:

* The exclusion criteria were neck pain that included inflammatory rheumatological diseases, malignancy, or structural deformity, previous surgery related to the cervical spine,
* Severe referred pain (greater than 7 on a 0-to-10 Visual Analogue Scale-VAS).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Postural Assessments | 5 minute
  Eye angle, craniovertebral angle,shoulder angle

SECONDARY OUTCOMES:
Performance | 10 minute
  6 minute walk test

OTHER OUTCOMES:
Energy Consumption | 15 minute
  Physiologic Cost Index

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Y Şahan, pHD, Study Director — University of Health science
Locations (1):
- Tezel Yıldırım Şahan, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Arshadi R, Ghasemi GA, Samadi H. Effects of an 8-week selective corrective exercises program on electromyography activity of scapular and neck muscles in persons with upper crossed syndrome: Randomized controlled trial. Phys Ther Sport. 2019 May;37:113-119. doi: 10.1016/j.ptsp.2019.03.008. Epub 2019 Mar 21. PMID 30928841
- [Background] Joshi S, Balthillaya G, Neelapala YVR. Thoracic Posture and Mobility in Mechanical Neck Pain Population: A Review of the Literature. Asian Spine J. 2019 Jun 3;13(5):849-860. doi: 10.31616/asj.2018.0302. Print 2019 Oct. PMID 31154701
- [Background] Hogg-Johnson S, van der Velde G, Carroll LJ, Holm LW, Cassidy JD, Guzman J, Cote P, Haldeman S, Ammendolia C, Carragee E, Hurwitz E, Nordin M, Peloso P. The burden and determinants of neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. J Manipulative Physiol Ther. 2009 Feb;32(2 Suppl):S46-60. doi: 10.1016/j.jmpt.2008.11.010. PMID 19251074
- [Background] Lohman EB, Pacheco GR, Gharibvand L, Daher N, Devore K, Bains G, AlAmeri M, Berk LS. The immediate effects of cervical spine manipulation on pain and biochemical markers in females with acute non-specific mechanical neck pain: a randomized clinical trial. J Man Manip Ther. 2019 Sep;27(4):186-196. doi: 10.1080/10669817.2018.1553696. Epub 2018 Dec 11. PMID 30935335
- [Background] de Araujo Cazotti L, Jones A, Roger-Silva D, Ribeiro LHC, Natour J. Effectiveness of the Pilates Method in the Treatment of Chronic Mechanical Neck Pain: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Sep;99(9):1740-1746. doi: 10.1016/j.apmr.2018.04.018. Epub 2018 May 9. PMID 29752907